CLINICAL TRIAL: NCT07348341
Title: Coronary Laser Atherectomy Registry From an International Taskforce
Acronym: CLARIT
Status: Not yet recruiting | Type: Observational
Sponsor: Ceric Sàrl (Industry)
Collaborators: Philips Medical Systems (Industry); European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: PHI-01
Record Dates: First submitted 2025-11-17; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stable Coronary Artery Disease; Acute Coronary Syndromes
Keywords: excimer laser coronary atherectomy; ELCA; CLARIT; coronary artery disease; acute coronary syndromes
MeSH Terms: conditions — Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Excimer Laser Coronary Atherectomy (ELCA) — ELCA treat a significant coronary stenosis or recanalize occluded coronary arteries using UV during percutaneous coronary intervention.

SUMMARY:
This study is a prospective, investigator-initiated, multi-center, single arm, observational registry of performance of Excimer Laser Coronary Atherectomy (ELCA) in standard use cases of percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
The primary objective of the CLARIT study is to assess the Safety and Efficacy of ELCA in recognized indications for the device at Index PCI and during the in-hospital stay. The secondary objectives includes the safety and efficacy of ELCA at 30 days and 1 year, as well as the procedural characteristics for the assessment of the learning curve and impact on the catheter lab workflow.

500 patients will be included in 20 sites accorss 8 countries in Europe, United Kingdom and India. The patients included in the study according to eligibility criteria will be followed up one year. The total study duration is 3 years, including 2 years of recruitment.

The follow-up/visit windows include the screening/baseline period, on the day of procedure, discharge; 1 month and 1 year follow-up. The ELCA is to be used following Instruction for uses and follow-up as per hospital standard of care.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if all the following criteria are met:

1. Age 18 years or over
2. Patient willing to be included in the registry
3. Patients with stable coronary artery disease or acute coronary syndromes with de-novo or intra-stent restenosis (ISR) coronary lesions suitable to be treated with ELCA

   * Non-Crossable with ICI catheter or:
   * Crossable with ICI catheter with significant calcium score suggesting need for calcium modification based on IVUS or OCT criteria and/or
   * Non-Dilatable with 1:1 NC balloon
4. Mandated use of ICI:

   * Attempted before use of ELCA or
   * Following ELCA and any other calcium modification strategy utilized (to evaluate whether the additional modification demonstrates significant additional modification of the calcium on ICI)
   * Final after DES implantation or prior to use of DCB
5. Declared PCI strategy (planned use of ELCA, need for IVL/specialty balloons/alternative atherectomy and stent strategy) prior to PCI procedure

Exclusion Criteria:

1. Pregnant or breast feeding
2. Unable to give informed consent
3. PCI performed without IVCI attempt
4. No ELCA use
5. Allergy to clopidogrel, prasugrel or ticagrelor or non-compliance
6. Post- cardiac arrest or haemodynamic instability
7. Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable coronary artery disease or acute coronary syndromes who will be treated with excimer laser coronary atherectomy (ELCA)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Procedural success during index PCI | During Procedure
  The primary endpoint of efficacy is procedural Success during index PCI:, which is a combined endpoint of these following events:
  * Angiographic success defined as residual stenosis <30% in two orthogonal projections after lesion treatment with ELCA destination therapy with DES or DCB
  * TIMI 3 flow and absence of ELCA related complications during the procedure
  * Intra-Coronary Imaging success defined as final MSA > 5.5mm2 IVUS or 4.5mm2 OCT with > 80% stent expansion - site reported
Freedom from in hospital Major Adverse Cardiovascular Events | Periprocedural
  The primary endpoint of safety is freedom from in-hospital Major Adverse Cardiovascular Events (MACE), including : cardiac death, target vessel myocardial infarction (TVMI), urgent repeat target vessel revascularization (TVR) with either PCI or CABG, and Stroke.

SECONDARY OUTCOMES:
Composite endpoint of one of events reported | 30 days and 1 year
  The secondary endpoint is a composite endpoint of one of these event : Major Adverse Cardiovascular Events (MACE) (including cardiac death, target vessel revascularization, myocardial infarction, target vessel myocardial infarction (TVMI), unplanned hospitalization of unstable angina).
Success of revascularization: Freedom from Target lesion failure (TLF) events and ICI assessed stent optimization | 30 days and 1 year
  This is defined by MSA stent expansion,stent apposition, full lesion coverage with < 50% plaque burden at proximal and distal references with TIMI 3 flow, no significant edge dissection
Procedural Characteristic- Cost | During procedure
  Procedural costs (devices used)
Procedural Characteristic- Device success based on maximum fluence | During procedure
  Device Success based on maximum fluence
Procedural Characteristic- Fluoroscopy Time | During procedure
  Fluoroscopy time
Procedural Characteristic- Contrast Volume | During procedure
  Contrast Volume
Procedural characteristic- Device success based on repetition rate | During procedure
  Device Success based on repetition rate
Procedural characteristic- Device success based on pulses number | During procedure
  Device Success based on number of pulses
Procedural characteristic- Device success based on lasing duration | During Procedure
  Device Success in relation to the duration of lasing
Procedural characteristic- Device success based on laser trains number | During procedure
  Device Success in relation to the number of laser trains
Procedural characteristic- Catheter access | During Procedure
  Catheter access : radial or femoral
Requirement of hemodynamic support | During procedure
  composite of need for pharmacological or mechanical hemodynamic support
Marker of the learning curve associated with ELCA- Total procedure time | During procedure
  The total time of the procedure
Marker of the learning curve associated with ELCA- Intra-procedural interval from ELCA decision to post-ELCA intracoronary imaging | During procedure
  The time between the decision for ELCA to the uses of Intracoronary imaging after ELCA.
Marker of the learning curve associated with ELCA- Number of ECLA trains | During procedure
  The number of ELCA trains, including the number of pulses, settings performed by the clinician.
Marker of the learning curve associated with ELCA- Milieu type used during lasing | During procedure
  The type of milieu used during lasing (blood, saline or contrast)
Impact on catheter lab workflow- Lesion preparation strategy | During procedure
  The change in lesion preparation strategy compared to the operator's initial upfront declared strategy (uses of IVL, specialty balloons or other atherectomy device alongside ELCA).
Impact on catheter lab workflow- Stent Strategy | During procedure
  The change of stent strategy (after ELCA and subsequent ICI) compared to the operator's initial upfront declared strategy.
Impact on catheter lab workflow- Procedural duration | During procedure
  Procedural duration for decision of ELCA to passage of Intracoronary imaging or ballon
Intracoronary imaging analysis by the site- Calcium morphology | During procedure
  Calcium morphology (concentric, eccentric or nodular) reported by the site.
Intracoronary imaging analysis by the site- Depth of lesion calcification | During procedure
  Depth of lesion calcification reported by the site.
Intracoronary imaging analysis by the site- Lesion calcification length | During procedure
  Length of lesion calcification reported by the site
Intracoronary imaging analysis by the CoreLab | During procedure
  calcium burden (%)
Intracoronary imaging analysis by the CoreLab | During Procedure
  calcium depth (mm)
Intracoronary imaging analysis by the CoreLab | During procedure
  impact of OAS and other devices on calcium
Intracoronary imaging analysis by the CoreLab | during procedure
  minimal stent area (mm²)
Intracoronary imaging analysis by the CoreLab | During Procedure
  stent expansion (%)
Intracoronary imaging analysis by the CoreLab | During Procedure
  presence of edge dissection
Intracoronary imaging analysis by the CoreLab | During procedure
  presence of stent malposition
Intracoronary imaging analysis by the CoreLab | During procedure
  maximal eccentricity index

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'kane, Professor, Study Chair — Dorset Heart Centre, The Royal Bournemouth Hospital

IPD SHARING:
Plan to Share IPD: Undecided